CLINICAL TRIAL: NCT05496881
Title: Evaluating Task-Oriented Exercise Effects on Walking Function and the Central Nervous System in People With Multiple Sclerosis
Brief Title: Exercise Effects in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regina (Other)
Collaborators: First Steps Wellness Centre (Unknown); Saskatchewan Health Research Foundation (Other); University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021-197
Record Dates: First submitted 2022-04-14; First posted 2022-08-11 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis
Keywords: Progressive Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Central Nervous System; Motor Learning; Transcranial Magnetic Stimulation; Mobility Limitation
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: All interventions will involve 60-minute sessions delivered three times per week for 12 weeks. All interventions will involve the whole body but differ in content.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be informed of the different study arms. Interventions will be scheduled to avoid contact between study arms. Participants will be asked to not describe their activities to those outside of their exercise group. Although it will not be possible to blind program instructors from the intervention that they deliver, instructors will not be aware of the expected results. Assessors and data analysts will be fully blinded to study arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Group 1 (Experimental): The intervention will focus on mobility and balance.
  Interventions: Other: Exercise Group 1
- Exercise Group 2 (Active Comparator): This intervention will focus on physical fitness.
  Interventions: Other: Exercise Group 2
- Exercise Group 3 (Sham Comparator): This intervention will focus on flexibility, range of motion, and muscle tone.
  Interventions: Other: Exercise Group 3

INTERVENTIONS:
Other: Exercise Group 1 — Prescribed exercises will focus on mobility and balance.
  Arms: Exercise Group 1
Other: Exercise Group 2 — Prescribed exercises will focus on physical fitness.
  Arms: Exercise Group 2
Other: Exercise Group 3 — Prescribed exercises will focus on flexibility, range of motion, and muscle tone.
  Arms: Exercise Group 3

SUMMARY:
A growing body of work suggests that regular exercise can support symptom management and improve physical function for people living with multiple sclerosis (MS). Although exercise is known to be beneficial for managing many symptoms related to MS, its effects on the central nervous system, and whether these effects change with different types of exercise, are not well understood. Here, the investigators have designed a clinical trial that compares the effects of distinct exercise protocols on aspects of physical function, physical fitness, and central nervous system function. This research will be the first to compare the effects of different types of exercise on central nervous system changes in people with MS.

DETAILED DESCRIPTION:
A total of 69 participants with multiple sclerosis (MS) and moderate motor disability in the province of Saskatchewan, Canada will be randomly assigned to receive one of three distinct exercise programs. All exercise programs will be delivered three times per week in 60-minute group sessions over the course of 12 weeks under the supervision of Clinical Exercise Physiologists. Exercise programming will include activities focused on mobility, fitness, and flexibility. Assessments of physical function, physical fitness, and central nervous system function will be conducted immediately before, after, and six weeks following completion of the exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of progressive MS by a neurologist
* physician clearance for exercise
* a Patient-Determined Disease Steps (PDSS) score between 3 and 7 (i.e., moderate motor disability)
* a Timed 25-Foot Walk (T25-FW) test time > 6.0 s.

Exclusion Criteria:

* a baseline score >24 on the Godin-Shephard Leisure Time Physical Activity Questionnaire (i.e., high physical activity levels)
* absolute contraindications to TMS (e.g. history of seizure)
* a history of any neurological conditions other than MS
* relapse in the past three months (self-reported, neurologist confirmed)
* psychiatric diagnosis
* substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Timed 25-Foot Walk Test | 6 weeks post intervention
  The Timed 25-Foot Walk Test provides an assessment of mobility and lower-extremity function through a measurement of fast walking speed. Test scores range from 0-180 seconds with higher values indicating a worse outcome.

SECONDARY OUTCOMES:
Motor Evoked Potential Amplitude | 6 weeks post intervention
  Measuring the amplitude of motor evoked potentials elicited by transcranial magnetic stimulation delivered over the motor cortex provides information about corticospinal excitability. Corticospinal excitability is a potential marker of MS disease burden that is responsive to physical training in people with MS and has been used to study experience-dependent neuroplasticity in other neurological conditions. The range of response amplitude is 0-100% of maximal muscle fibre recruitment, with higher values indicating better outcome.

OTHER OUTCOMES:
Mini Balance Evaluation Systems Test | 6 weeks post intervention
  The Mini Balance Evaluation Systems Test provides an assessment of balance control systems. The Mini-BESTest has a high sensitivity in detecting balance impairments in people with MS. The Mini-BESTest has score values between 0-28 with a higher score meaning a better outcome.
Multiple Sclerosis Impact Scale | 6 weeks post intervention
  The Multiple Sclerosis Impact Scale is a self-report survey that measures the impact of multiple sclerosis on physical and psychological functioning. The MSIS test has a score value between 0-145 with a higher score meaning a worse outcome.
9-Hole Pegboard Test | 6 weeks post intervention
  The 9-Hole Pegboard Test is a quantitative measure of upper extremity function. The test has a time limit of 300 seconds with higher values indicating a worse outcome.
Symbol Digit Modalities Test | 6 weeks post intervention
  The Symbol Digit Modalities Test is used to asses divided attention, visual scanning, tracking and motor speed. The SDMT test is scored as the number of correct answers provided within 90 seconds (range: 0-110). A higher score would indicate a better outcome.
Peak Isometric Hand Grip Force | 6 weeks post intervention
  Peak Isometric Hand Grip Force provides a measure of general upper-extremity strength. Values typically range from 0 to approximately 75 kilograms of force, with higher values indicating greater strength.
Peak Isometric Knee Extensor Torque | 6 weeks post intervention
  Peak Isometric Knee Extensor Torque provides a measure of general lower-extremity strength. Values typically range from 0 to approximately 75 kg of force, with higher values indicating greater strength. Values typically range from 0 to approximately 300 Newton*Meters of torque, with higher values indicating greater strength.
Peak Oxygen Uptake | 6 weeks post intervention
  Peak Oxygen Uptake provides a measure of cardiorespiratory fitness. It is measured through administration of a maximal exercise test. Values typically range from 0-90 milliliters per minute per kilogram.
Tumor Necrosis Factor Alpha concentration in systemic blood | 6 weeks post intervention
  Tumor Necrosis Factor is an inflammatory cytokine that can be measured in human blood serum. Values typically range from 100 to 5000 picograms per milliliter of blood serum. Higher values are generally considered worse.
Brain-Derived Neurotrophic Factor in systemic blood | 6 weeks post intervention
  Brain-Derived Neurotrophic Factor is a neurotrophic growth factor that can be measured in human blood serum. Values typically range from 15 to 80 nanograms per milliliter of blood serum. Higher values are generally considered better.
Neurofilament Light concentration in systemic blood | 6 weeks post intervention
  Neurofilament Light is a neuronal cytoplasmic protein that can be measured in human blood serum. Values typically range from 0 to 100 picograms per milliliter of blood serum. Higher values are generally considered worse.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Mang, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

REFERENCES:
- [Background] Warraich Z, Kleim JA. Neural plasticity: the biological substrate for neurorehabilitation. PM R. 2010 Dec;2(12 Suppl 2):S208-19. doi: 10.1016/j.pmrj.2010.10.016. PMID 21172683
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Background] Goldman MD, Motl RW, Scagnelli J, Pula JH, Sosnoff JJ, Cadavid D. Clinically meaningful performance benchmarks in MS: timed 25-foot walk and the real world. Neurology. 2013 Nov 19;81(21):1856-63. doi: 10.1212/01.wnl.0000436065.97642.d2. Epub 2013 Oct 30. PMID 24174581
- [Background] Chaves AR, Devasahayam AJ, Kelly LP, Pretty RW, Ploughman M. Exercise-Induced Brain Excitability Changes in Progressive Multiple Sclerosis: A Pilot Study. J Neurol Phys Ther. 2020 Apr;44(2):132-144. doi: 10.1097/NPT.0000000000000308. PMID 32168157
- [Background] Snow NJ, Wadden KP, Chaves AR, Ploughman M. Transcranial Magnetic Stimulation as a Potential Biomarker in Multiple Sclerosis: A Systematic Review with Recommendations for Future Research. Neural Plast. 2019 Sep 16;2019:6430596. doi: 10.1155/2019/6430596. eCollection 2019. PMID 31636661
- [Background] Kieseier BC, Pozzilli C. Assessing walking disability in multiple sclerosis. Mult Scler. 2012 Jul;18(7):914-24. doi: 10.1177/1352458512444498. Epub 2012 Apr 24. PMID 22740603
- [Background] Phan-Ba R, Pace A, Calay P, Grodent P, Douchamps F, Hyde R, Hotermans C, Delvaux V, Hansen I, Moonen G, Belachew S. Comparison of the timed 25-foot and the 100-meter walk as performance measures in multiple sclerosis. Neurorehabil Neural Repair. 2011 Sep;25(7):672-9. doi: 10.1177/1545968310397204. Epub 2011 Mar 24. PMID 21436388
- [Background] Coleman CI, Sobieraj DM, Marinucci LN. Minimally important clinical difference of the Timed 25-Foot Walk Test: results from a randomized controlled trial in patients with multiple sclerosis. Curr Med Res Opin. 2012 Jan;28(1):49-56. doi: 10.1185/03007995.2011.639752. Epub 2011 Nov 23. PMID 22073939
- [Background] Motl RW, Cohen JA, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the timed 25-foot walk as an ambulatory performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):704-710. doi: 10.1177/1352458517690823. Epub 2017 Feb 16. PMID 28206828
- [Background] Yen CL, Wang RY, Liao KK, Huang CC, Yang YR. Gait training induced change in corticomotor excitability in patients with chronic stroke. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):22-30. doi: 10.1177/1545968307301875. Epub 2007 May 16. PMID 17507641
- [Background] Guerra E, di Cagno A, Mancini P, Sperandii F, Quaranta F, Ciminelli E, Fagnani F, Giombini A, Pigozzi F. Physical fitness assessment in multiple sclerosis patients: a controlled study. Res Dev Disabil. 2014 Oct;35(10):2527-33. doi: 10.1016/j.ridd.2014.06.013. Epub 2014 Jul 5. PMID 25000308
- [Background] Pilutti LA, Sandroff BM, Klaren RE, Learmonth YC, Platta ME, Hubbard EA, Stratton M, Motl RW. Physical Fitness Assessment Across the Disability Spectrum in Persons With Multiple Sclerosis: A Comparison of Testing Modalities. J Neurol Phys Ther. 2015 Oct;39(4):241-9. doi: 10.1097/NPT.0000000000000099. PMID 26247510
- [Derived] Moslemi Z, Toledo-Aldana EA, Baldwin B, Donkers SJ, Eng JJ, Mondal P, de Zepetnek JOT, Buttigieg J, Levin MC, Mang CS. Task-oriented exercise effects on walking and corticospinal excitability in multiple sclerosis: protocol for a randomized controlled trial. BMC Sports Sci Med Rehabil. 2023 Dec 21;15(1):175. doi: 10.1186/s13102-023-00790-5. PMID 38129896